CLINICAL TRIAL: NCT02129400
Title: Xenon-inhalation: Elimination of Xenon and Its Effect on Erythropoetin Levels in Blood of Healthy Volunteers
Brief Title: Influence on Erythropoetin-level by Xenon
Acronym: XEPO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The analysis of the blood samples was much expensive than calculated. The recruitment had to be stopped after 36 study participants.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-026; 2014-000973-38 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-05-02 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Xenon-inhalation; Erythropoetin; Pharmakokinetic; Pharmacodynamic; Hemodynamic parameters; Inflammatory parameters; Growth factors; Oxidative stress parameters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- 10min Xenon 15%, FiO2 75% (Experimental): 10 minutes of 15 % xenon-inhalation (with 75 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 10min Xenon 30%, FiO2 60% (Experimental): 10 minutes of 30 % xenon-inhalation (with 60 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 30min Xenon 15%, FiO2 75% (Experimental): 30 minutes of 15 % xenon-inhalation (with 75 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 30min Xenon 30%, FiO2 60% (Experimental): 30 minutes of 30 % xenon-inhalation (with 60 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 45min Xenon 15%, FiO2 75% (Experimental): 45 minutes of 15 % xenon-inhalation (with 75 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 45min Xenon 30%, FiO2 60% (Experimental): 45 minutes of 30 % xenon-inhalation (with 60 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 90min Xenon 15%, FiO2 75% (Experimental): 90 minutes of 15 % xenon-inhalation (with 75 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 90min Xenon 30%, FiO2 60% (Experimental): 90 minutes of 30 % xenon-inhalation (with 60 % FiO2)
  Interventions: Drug: Xenon pro Anaesthesia 100 % (V/V)
- 10min air medicinalis, FiO2 75% (Placebo Comparator): 10 minutes of air medicinalis (with 75 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 10min air medicinalis, FiO2 60% (Placebo Comparator): 10 minutes of air medicinalis inhalation (with 60 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 30min air medicinalis, FiO2 75% (Placebo Comparator): 30 minutes of air medicinalis inhalation (with 75 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 30min air medicinalis, FiO2 60% (Placebo Comparator): 30 minutes of air medicinalis inhalation (with 60 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 45min air medicinalis, FiO2 75% (Placebo Comparator): 45 minutes of air medicinalis inhalation (with 75 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 45min air medicinalis, FiO2 60% (Placebo Comparator): 45 minutes of air medicinalis inhalation (with 60 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 90min air medicinalis, FiO2 75% (Placebo Comparator): 90 minutes of air medicinalis inhalation (with 75 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%
- 90min air medicinalis, FiO2 60% (Placebo Comparator): 90 minutes of air medicinalis inhalation (with 60 % FiO2)
  Interventions: Drug: Aer medicinalis Linde 100%

INTERVENTIONS:
Drug: Xenon pro Anaesthesia 100 % (V/V) — Xenon-gas inhalation of indicated concentrations during indicated time
  Other Names: licence number: 56582.00.00
  Arms: 10min Xenon 15%, FiO2 75%; 10min Xenon 30%, FiO2 60%; 30min Xenon 15%, FiO2 75%; 30min Xenon 30%, FiO2 60%; 45min Xenon 15%, FiO2 75%; 45min Xenon 30%, FiO2 60%; 90min Xenon 15%, FiO2 75%; 90min Xenon 30%, FiO2 60%
Drug: Aer medicinalis Linde 100%
  Other Names: Pharmakotherapeutic group: medical gas; Licence number: 68885.00.00; ATC-Code: V03AN05
  Arms: 10min air medicinalis, FiO2 60%; 10min air medicinalis, FiO2 75%; 30min air medicinalis, FiO2 60%; 30min air medicinalis, FiO2 75%; 45min air medicinalis, FiO2 60%; 45min air medicinalis, FiO2 75%; 90min air medicinalis, FiO2 60%; 90min air medicinalis, FiO2 75%

SUMMARY:
The purpose of this study is to analyze the effect of xenon-inhalation on erythropoetin-level in blood of healthy volunteers and to determine the efficient time of inhalation.

Hypothesis: Xenon-inhalation enhances erythropoetin-levels in blood

DETAILED DESCRIPTION:
Xenon-gas is an approved anesthetic by the EMEA and is used for a balanced anesthesia in combination with opioids for adults with a american society of anesthesiology classification ASA ≤ III. Several clinical and pre-clinical studies have shown a positive effect of xenon on several organ functions such as in brain, kidneys and heart. In two studies, an enhanced expression of hypoxia inducible factor-1α (HIF-1α) could be shown in animal kidneys and kidney cells. Interestingly, HIF-1α leads to an enhanced formation of erythropoetin (EPO). This might result in an enhanced oxygen transport capacity and an enhanced oxygen-level after xenon-treatment.

Aim of the project is to analyze the effect of xenon-inhalation on circulating erythropoetin-level in blood of healthy volunteers in a randomized controlled pilot study. Besides, other positive stimulating factors for erythropoiesis (such as HIFa stabilizing factors) and growth factors (such as fibroblast growth factors (FGFs), hepatocyte growth factor (HGF), mechano growth factors (MGFs), platelet-derived growth factors (PDGFs), vascular endothelial growth factors (VEGFs)) shall be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Age: > 18 years
* legally competent to sign
* without any known medical condition or medication prescribed at the University Hospital RWTH Aachen, Germany
* Persons that are able and willing to understand and follow the instructions of the study personnel
* Signed informed consent

Exclusion Criteria:

* Smoker, alcoholic or person who regularly consumes drugs or medication
* Persons with a medical condition that is contraindicated with the planned treatment
* Known hypersensitivity against xenon
* Persons not legally competent to sign
* Simultaneous participation at any other trial
* Blood-loss due to trauma during the period of the study or 2 months previous
* Blood donation during the period of the study or 2 months previous

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in erythropoetin-level in blood of healthy volunteers up to 216 hrs after the first of three xenon applications in total | up to 216 hrs after first xenon-application
  Change from baseline in erythropoetin-level in blood of healthy volunteers up to 216 hrs after the first of three xenon applications in total.
  Timepoints of measurement:
  Before each inhalation, Directly after the first inhalation, 2 hrs after the first inhalation, 4 hrs after the first inhalation, 8 hrs after the first inhalation, 22-24 hrs after each inhalation, 46-48 hrs after each inhalation, 70-72 hrs after the last inhalation, 94-96 hrs after the last inhalation, 118-120 hrs after the last inhalation

SECONDARY OUTCOMES:
First-order elimination of xenon after xenon-inhalation in blood and exhalation air by mass-spectroscopy | up to 216 hrs after the first xenon-application
  Timepoints of measurement:
  Before each inhalation, Directly after the first inhalation, 2 hrs after the first inhalation, 4 hrs after the first inhalation, 8 hrs after the first inhalation, 22-24 hrs after each inhalation, 46-48 hrs after each inhalation, 70-72 hrs after the last inhalation, 94-96 hrs after the last inhalation, 118-120 hrs after the last inhalation

OTHER OUTCOMES:
Determination of hemodynamic parameters (HF, RR, EKG, SpO2, rSO2, tSO2) | up to 216 hrs after the first xenon-application
  Time points of measurement:
  Before each inhalation, Directly after the first inhalation, 2 hrs after the first inhalation, 4 hrs after the first inhalation, 8 hrs after the first inhalation, 22-24 hrs after each inhalation, 46-48 hrs after each inhalation, 70-72 hrs after the last inhalation, 94-96 hrs after the last inhalation, 118-120 hrs after the last inhalation
Laboratory parameters: Inflammation (procalcitonin, IL-6, IL-10, leukocytes, thrombocytes), growth factors (HIF1α, FGFs, HGF, MGFs, PDGF, VEGF, IL-8, VEGF, MIF, SDF-1a) | up to 216 hrs after the first xenon-application
  Timepoints of measurement:
  Before each inhalation, Directly after the first inhalation, 2 hrs after the first inhalation, 4 hrs after the first inhalation, 8 hrs after the first inhalation, 22-24 hrs after each inhalation, 46-48 hrs after each inhalation, 70-72 hrs after the last inhalation, 94-96 hrs after the last inhalation, 118-120 hrs after the last inhalation
Oxidative stress: total oxidative capacity, peroxide activity, LDL antibodies: antibody against oxided LDL, e.g. MDA-LDL IgM, oLAb (IgG) | up to 216 hrs after the first xenon-application
  Time points of measurement:
  Before each inhalation, Directly after the first inhalation, 2 hrs after the first inhalation, 4 hrs after the first inhalation, 8 hrs after the first inhalation, 22-24 hrs after each inhalation, 46-48 hrs after each inhalation, 70-72 hrs after the last inhalation, 94-96 hrs after the last inhalation, 118-120 hrs after the last inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. M.D., Principal Investigator — University Hospital RWTH Aachen, Department for Anesthesia
Locations (1):
- University Hospital RWTH Aachen, Department for Anesthesia, Aachen, North-Rhine Westfalia, Germany